CLINICAL TRIAL: NCT04525651
Title: Clinical Evaluation for Digital Acupuncture Manipulation Therapeutic Instrument
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: lhzj20200810
Record Dates: First submitted 2020-08-11; First posted 2020-08-25 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Cervical Spondylosis
Keywords: digital acupuncture manipulation therapeutic instrument; cervical spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Acupuncture Instrument Group (Experimental): The needles will be stimulated manually to achieve de qi (a compositional sensation including soreness, numbness, distention and heaviness) and then paired electrodes from the digital acupuncture instrument will be attached to the needle handles and another two adjunct acupoints by the research assistant. The electric current will be increased until the needles begin to vibrate slightly.
  Interventions: Device: Digital Acupuncture Manipulation Therapeutic Instrument
- Manual Acupuncture Group (Active Comparator): Patients in the MA group will undergo similar procedures as the EA group except that no current will be output from the instrument.
  Interventions: Other: Manual Acupuncture
- Sham Acupuncture Group (Sham Comparator): Patients in the SA group will receive non-invasive acupuncture to avoid de qi.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Device: Digital Acupuncture Manipulation Therapeutic Instrument — The device is based on the characteristics of traditional acupuncture manipulation of Shanghai School of Traditional Chinese Medicine, and absorbs the information of the techniques of famous experts, modulates the stimulation waveform of the electroacupuncture device by modulating the signal, and realizes the digitization of acupuncture technique information.
  Arms: Digital Acupuncture Instrument Group
Other: Manual Acupuncture — Manual acupuncture to acheive de qi.
  Arms: Manual Acupuncture Group
Other: Sham Acupuncture — Sham acupuncture to avoid de qi.
  Arms: Sham Acupuncture Group

SUMMARY:
The investigators design a randomized, control study to evaluate the therapeutic effect of digital acupuncture instrument in cervical spondylotic radiculopathy patients using the following outcomes: the Visual analogue scale(VAS), neck disability index scale (NDI) and short form 36-item questionnaire (SF-36).

DETAILED DESCRIPTION:
Based on the digital acupuncture manipulation therapeutic instrument developed in the previous stage, the acupuncture manipulation acquisition system is used to compare and analyze the analog waves output by the experts' acupuncture manipulation and the manipulative therapeutic apparatus in the system data analysis module, in order to verify the consistency of bioelectric signals of different reinforcing and reducing manipulation of acupuncture and experts' manipulation. The biocompatibility of shock wave was detected by Massachusetts General Hospital Needle sensation scale ((Massachusetts General Hospital Acupuncture Sensation Scale, MASS)). The visual analogue pain score ((Visual analogue scale, VAS)), neck disability index scale ((Neck Disability Index,NDI) and short form 36-item questionnaire (SF-36) were used to evaluate the clinical efficacy and safety of the instrument in the treatment of cervical pain in cervical Spondylotic radiculopathy, and the appropriate syndrome type of the scheme was studied.

ELIGIBILITY:
Inclusion Criteria:

1. Neck pain with the diagnosis of cervical spondylotic radiculopathy;
2. Aged between 18-70 years;
3. Have not participated in any drug clinical trials within the last month;
4. Voluntarily joining this study with informed consents

Exclusion Criteria:

1. A history of cervical spine trauma or have received cervical spine surgery;
2. Accompanied by obvious dizziness and spinal cord compression symptoms or imaging findings of spinal cord compression;
3. Cervical spondylosis in urgent need of surgery;
4. Pregnant women and lactating women;
5. A serious heart condition, hepatic disease, renal system disease, hematopoietic system disease, or whole-body malnutrition
6. Anticoagulant treatments such as warfarin or heparin use of pacemakers or receiving acupuncture in the past 2 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale（VAS） | Change from baseline VAS at 4weeks
  A graphic scale that helps a patient to quantify pain, depression, and other subjective and otherwise unmeasurable states or conditions.
Visual Analogue scale（VAS） | Change from baseline VAS at 8weeks
  A graphic scale that helps a patient to quantify pain, depression, and other subjective and otherwise unmeasurable states or conditions.

SECONDARY OUTCOMES:
Neck Disability Index（NDI） | Baseline(Week 0), After treatment(Week 4), Follow-up(Week 8)
  A scale that helps a patient to quantify neck disability.
short form 36-item questionnaire, SF-36 | Baseline(Week 0), After treatment(Week 4), Follow-up(Week 8)
  a set of 36 questions abstracted from the much longer set of several hundred used in household interview surveys of the U.S. National Health Survey. The SF36 questions are a convenient abbreviation, used for screening purposes to assess the physical function, social function, role limitation, mental health, energy, vitality, pain, and subjective perception of health status. They have been tested and found to be valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, Doctor, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- LongHua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China